CLINICAL TRIAL: NCT04981223
Title: Predicting Location and Extent of Prostate Cancer Using Micro-Ultrasound Imaging
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Geoffrey Sonn, Associate Professor of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-58101; NCI-2022-05158 (Registry Identifier: National Cancer Institute: Clinical Trials Reporting Program)
Record Dates: First submitted 2021-07-09; First posted 2021-07-28 (Actual); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ExactVu Imaging (Experimental): EV29L transducer will be inserted in the subject's rectum. Cine sweeps will be performed to save images of:
  1. The entire prostate from posterior to anterior (may require 2 sweeps to cover base and apex)
  2. The peripheral zone using the highest zoom setting (30mm depth) on the system (may require 2 sweeps to cover base and apex). Analysis of these images will be performed after surgery but before prostatectomy
  Interventions: Device: ExactVu

INTERVENTIONS:
Device: ExactVu — clinical micro-ultrasound, imaging Device, Manufacturer; Exact Imaging

SUMMARY:
The goal of this study is to use a clinical micro-ultrasound to systematically image the prostate before biopsy or surgery. The images from the ultrasound system will be saved and compared to other imaging modalities and pathology in order to develop better tools.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for MR-US fusion prostate biopsy or radical prostatectomy
* Agree to consent to the study

Exclusion Criteria:

* Does not agree to consent.

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Sonn, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou SR, Choi MH, Vesal S, Kinnaird A, Brisbane WG, Lughezzani G, Maffei D, Fasulo V, Albers P, Zhang L, Kornberg Z, Fan RE, Shao W, Rusu M, Sonn GA. Inter-reader Agreement for Prostate Cancer Detection Using Micro-ultrasound: A Multi-institutional Study. Eur Urol Open Sci. 2024 Jul 13;66:93-100. doi: 10.1016/j.euros.2024.06.017. eCollection 2024 Aug. PMID 39076245

RESULTS

PARTICIPANT FLOW:
Groups:
- ExactVu Imaging: EV29L transducer will be inserted in the subject's rectum. Cine sweeps will be performed to save images of:
  1. The entire prostate from posterior to anterior (may require 2 sweeps to cover base and apex)
  2. The peripheral zone using the highest zoom setting (30mm depth) on the system (may require 2 sweeps to cover base and apex). Analysis of these images will be performed after surgery but before prostatectomy
  ExactVu: clinical micro-ultrasound, imaging Device, Manufacturer; Exact Imaging
Period: Overall Study
Arm/Group | ExactVu Imaging
Started | 95
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ExactVu Imaging
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 85
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 62
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Micro-Ultrasound Detection of High Grade Prostate Cancer (Gleason Score ≥7) vs. Surgical Pathology
Description: Evaluate the ability of micro-ultrasound to identify high grade prostate cancer foci (Gleason score ≥7) in comparison to final surgical pathology result (prostatectomy or biopsy)
Time Frame: From date of micro ultrasound exam until the date of Prostate biopsy data are obtained (average of 7 days)
Measure: Number; unit: participants
Arm/Group | ExactVu Imaging
Number analyzed (Participants) | 57
participants
  Sensitivity (All Lesions) | 38
  Sensitivity (Excluding Anterior Lesions) | 50

2. Secondary Outcome: Prostate Cancer Border Identification Post-Prostatectomy
Description: Evaluate the ability of micro-ultrasound to identify the borders of prostate cancer foci in comparison to final surgical pathology result in men after prostatectomy.
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Micro-Ultrasound Detection of Low Grade Prostate Cancer (Gleason Score 6)
Description: Evaluate the ability of micro-ultrasound to detect low grade prostate cancer foci (Gleason score 6)
Time Frame: 1 year and 10 months
Measure: Number; unit: percentage of agreement
Arm/Group | ExactVu Imaging
Number analyzed (Participants) | 57
percentage of agreement
  Inter-Reader Agreement | 22
  Positive Percent Agreement for Low-Grade Cancers (Gleason Score 6) | 25.5

4. Secondary Outcome: Prostate Cancer Detection: Micro-Ultrasound vs. mpMRI Comparison
Description: Comparison of prostate cancer detection between micro-ultrasound and multiparametric magnetic resonance imaging (mpMRI).
Time Frame: 1 year and 10 months
Population: This analysis includes all participants evaluated for prostate cancer detection using micro-ultrasound (MUS) and multiparametric MRI (mpMRI). Metrics include sensitivity and inter-reader agreement (κ values), reported as percentages for consistency
Measure: Mean (Standard Error); unit: percentage of agreement
Arm/Group | ExactVu Imaging
Number analyzed (Participants) | 57
percentage of agreement
  Average Micro-Ultrasound Sensitivity | 66 (6.25)
  Average mpMRI Sensitivity | 90 (3.97)
  Average Micro-Ultrasound Inter-Reader Agreement (κ) | 30 (6.08)
  Average mpMRI Inter-Reader Agreement (κ) | 50 (6.63)

5. Secondary Outcome: Measuring Correlation Between Prostatectomy Pathology and Imaging Correlation
Description: Perform a detailed pathologic and imaging correlation between findings on micro-ultrasound, MRI and final surgical histopathology in men who undergo prostatectomy
Time Frame: 3 years
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: up to 3 months
Arm/Group | ExactVu Imaging
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT04981223/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04981223/ICF_000.pdf